CLINICAL TRIAL: NCT03886454
Title: Incidence and Nature of Respiratory Impairment in Consecutive Patients Undergoing Bronchoscopy Under Conscious Sedation: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: Natalie V. Zucker Research Grant (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB # 12489
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Conscious Sedation; Bronchoscopy
Keywords: Central apnea; Obstructive apnea; Oxygen desaturation; Escalation of Care; conscious sedation; Bronchoscopy; Respiratory impairment
MeSH Terms: conditions — Sleep Apnea, Central; Sleep Apnea, Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

SUMMARY:
This study aims to characterize airflow patterns during bronchoscopy under conscious sedation, and determine the incidence of obstructive and central respiratory events. The investigators also plan to monitor the degree and frequency of oxygen desaturation throughout the procedure. To achieve this, investigators use a physiologic monitoring device (NOX T3, K082113) that has been FDA approved for the screening and diagnosis of sleep disordered breathing [1]. The results from this pilot study will be used to assess the feasibility of a prospective study utilizing continuous external negative pressure (Pneuway). This negative pressure is applied through a neck mask to alleviate upper airway collapsibility and can potentially decrease the number of apneas during bronchoscopy under conscious sedation [2].

DETAILED DESCRIPTION:
Background and Rationale:

Diagnostic bronchoscopic procedures are commonly performed in patients with various forms of pulmonary disorders associated with abnormal chest imaging. During these procedures, the vocal cords are intubated using a flexible scope. Patients need sedation and analgesia, and conscious sedation is typically administered. Hypoxemia is a potential complication during bronchoscopy. Contributing factors in addition to the underlying lung pathology, include depression of the respiratory center and decreased upper airway muscle tone that occur during conscious sedation [3]. Upper airway obstruction including obstructive apnea is often unrecognized during these procedures till hypoxemia is apparent [4]. Propofol, a common drug used for conscious sedation, is known to cause respiratory depression, and potentially central and/or obstructive apneas with a direct dose-response pattern [5]. Others, including benzodiazepines and opiates, can also cause respiratory depression leading to central or obstructive events. Respiratory depression is potentiated when any of the above medications are combined [6].

Objectives:

The objective of the study is to identify the incidence of airflow limitation during bronchoscopy under conscious sedation, and further characterize it as obstructive or central. The primary endpoint is the incidence of obstructive and central apneic events during bronchoscopic procedures. The secondary outcomes include incidence of oxygen desaturation and need for escalation of care.

Study Design:

After informed consent is obtained, the NOX-T3 monitoring system, a commonly used portable sleep device that detects obstructive and central apneas, is placed prior to starting the procedure, and remains in place up to 30 minutes following the procedure. The NOX-T3 monitoring system includes a nasal cannula that sits over the nares, an elastic band that goes around the chest, and another one that goes around the abdomen, and a finger probe that is placed on the index finger. All subjects undergo bronchoscopy with standard of care including the monitoring of blood pressure, respiratory rate and oxygen saturation. All subjects have the NOX-T3 applied in addition to standard of care monitoring. Data is assessed following the completion of the procedure. Subjects' participation in this study ends at the completion of their standard of care visit. All the NOX-T3 studies are scored and interpreted by study investigators.

Data Management:

This is an observational and descriptive study with an estimated sample size of 30. Data collected will be reviewed with a statistician and investigators will report on patients' demographics. The study investigators will also present the incidence of apneic respiratory events and characterize them as obstructive or centrals. Investigators will further differentiate obstructive respiratory events to either apneas or hypopnea. Data on oxygen desaturations unrelated to apneic events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with respiratory pathology that require bronchoscopy for further diagnostic evaluation, as part of standard of care
2. Age of 18 years or older.
3. Our study does not include the recruitment of vulnerable populations such as cognitively impaired adults, pregnant women, pregnant minors, minors, wards of the state, non-viable neonates, neonates of uncertain viability and prisoners.

Exclusion Criteria:

1. Oxygen requirement of more than 4 Liter prior to procedure.
2. Intubation or any airway support.
3. Presence of severe cardiopulmonary or neurologic disease as determined by the investigator.
4. Nasal congestion/obstruction preventing proper placement and monitoring of air flow
5. Inability to provide informed consent.
6. All vulnerable population mentioned above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have been referred to the pulmonary division at Tufts Medical Center for bronchoscopy
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The incidence of obstructive and central apneic events. | Throughout the bronchoscopic procedure.
  Obstructive apnea are defined as more than 90% cessation of air-flow that lasts for at least 10 seconds, despite the presence of respiratory and abdominal muscle effort. Obstructive hypopnea is when more than 30% cessation of air-flow occurs that lasts for at least 10 seconds, and is associated with oxygen desaturation of at least 3% from baseline. Central apnea is when cessation of air-flow occurs secondary to absent respiratory and abdominal muscle effort, that lasts for at least 10 seconds.

SECONDARY OUTCOMES:
Oxygen desaturation | Throughout the bronchoscopic procedure.
  Oxygen desaturation of more than 3% from baseline which are unrelated to apneic events.
Need for escalation of care | Throughout the bronchoscopic procedure.
  Need for escalation of care, including but not limited to, increasing supplemental oxygen, jaw thrust, patient stimulation or interrupting the administration of conscious sedation drug.

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Ismail, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make IPD available to sommetrics Inc. to review once the study is complete. Data would include all the information obtained on the NOX-T3 device during conscious sedation which includes, but is not limited to, heart rate, respiratory rate, air flow through nasal cannula, oxygen saturation and chest and abdominal wall movements.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will become available after completion of the study and will be available to review for 1 year thereafter.
Access Criteria: IPD that is acquired by the NOX-T3 device is transferred to NOX-T3 software. Plan is to share IPD with sommetrics Inc. via that software.

REFERENCES:
- [Background] Cairns A, Wickwire E, Schaefer E, Nyanjom D. A pilot validation study for the NOX T3(TM) portable monitor for the detection of OSA. Sleep Breath. 2014 Sep;18(3):609-14. doi: 10.1007/s11325-013-0924-2. Epub 2014 Jan 19. PMID 24442914
- [Background] Kais SS, Klein KB, Rose RM, Endemann S, Coyle WJ. Continuous negative external pressure (cNEP) reduces respiratory impairment during screening colonoscopy: a pilot study. Endoscopy. 2016 Jun;48(6):584-7. doi: 10.1055/s-0042-102533. Epub 2016 Apr 25. PMID 27110692
- [Background] Hillman DR, Platt PR, Eastwood PR. The upper airway during anaesthesia. Br J Anaesth. 2003 Jul;91(1):31-9. doi: 10.1093/bja/aeg126. PMID 12821563
- [Background] Vargo JJ, Zuccaro G Jr, Dumot JA, Conwell DL, Morrow JB, Shay SS. Automated graphic assessment of respiratory activity is superior to pulse oximetry and visual assessment for the detection of early respiratory depression during therapeutic upper endoscopy. Gastrointest Endosc. 2002 Jun;55(7):826-31. doi: 10.1067/mge.2002.124208. PMID 12024135
- [Background] Eastwood PR, Platt PR, Shepherd K, Maddison K, Hillman DR. Collapsibility of the upper airway at different concentrations of propofol anesthesia. Anesthesiology. 2005 Sep;103(3):470-7. doi: 10.1097/00000542-200509000-00007. PMID 16129969
- [Background] Jose RJ, Shaefi S, Navani N. Sedation for flexible bronchoscopy: current and emerging evidence. Eur Respir Rev. 2013 Jun 1;22(128):106-16. doi: 10.1183/09059180.00006412. PMID 23728864